CLINICAL TRIAL: NCT01234181
Title: Clinical Study of Hypoxia-Stressed Bone Marrow Mononuclear Cell Intracoronary Transplantation in Myocardial Infarction and Other Heart Diseases.
Brief Title: Clinical Study of Hypoxia-Stressed Bone Marrow Mononuclear Cell Transplantation to Treat Heart Diseases
Acronym: CSHSBMMCTTHD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Jian'an Wang / Director, Chief of Heart Center, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAHZJU CT001; SFDA2010 (Registry Identifier: State Food and Drug Administration)
Record Dates: First submitted 2010-11-03; First posted 2010-11-04 (Estimated); Last update posted 2010-11-04 (Estimated); Status verified 2010-11

CONDITIONS: Myocardial Infarction (MI) or Acute Myocardial Infarction (AMI)
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BMSCs transplantation (Experimental)
  Interventions: Procedure: Hypoxia-stressed BMSCs transplantation to cure MI
- No BMSCs transplantation (Sham Comparator)
  Interventions: Procedure: Hypoxia-stressed BMSCs transplantation to cure MI

INTERVENTIONS:
Procedure: Hypoxia-stressed BMSCs transplantation to cure MI — Experimental group: intracoronary injection of 10^7 BMSCs Sham Comparator: inject the same volume saline

SUMMARY:
The purpose of this study, is to determine the differences of clinical outcomes between hypoxic pre-treatment group and control group in bone marrow stem cell transplantation (BM-SCT) to treat acute myocardial infarction (AMI); and to evaluate the safety of both treatments. Heart failure patients underwent PCI treatment after AMI and with informed consent, are randomized allocation into hypoxic pre-treated BM-SCT group, normoxic pre-treated BM-SCT group, and control group. Cell resuspension is intracoronary injected into patients receiving coronary angiography, IL-6, CRP, TNF and BNP are detected; echocardiography, cardiac MRI and ECT are analyzed to evaluate heart function and alive myocardial cells. Holter's ECG monitor is employed to observe arrhythmia and embolism. We hypothesize that, by receiving hypoxic pre-treated BM-SCT, impaired heart function will be reversed in heart failure patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute Myocardial Infarction(within one month);
* Age under 65;
* Infarction related wall motion abnormality on echocardiography;
* Infarction related TIMI flow grades 3 on coronary angiography during cell injection;
* Informed consent;

Exclusion Criteria:

* Active infection, or hematopoietic malignancy;
* Patients have tumor or other lethal diseases;
* Informed refusal

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-11; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Heart function | one year

CONTACTS AND LOCATIONS:
Overall Officials: Jian'an Wang, M.D, Ph.D, Principal Investigator — 2nd Affiliated Hospital, School of Medicine at Zhejiang University

REFERENCES:
- [Background] Hu X, Yu SP, Fraser JL, Lu Z, Ogle ME, Wang JA, Wei L. Transplantation of hypoxia-preconditioned mesenchymal stem cells improves infarcted heart function via enhanced survival of implanted cells and angiogenesis. J Thorac Cardiovasc Surg. 2008 Apr;135(4):799-808. doi: 10.1016/j.jtcvs.2007.07.071. PMID 18374759
- [Derived] Hu X, Huang X, Yang Q, Wang L, Sun J, Zhan H, Lin J, Pu Z, Jiang J, Sun Y, Xiang M, Liu X, Xie X, Yu X, Chen Z, Tse HF, Zhang J, Wang J. Safety and efficacy of intracoronary hypoxia-preconditioned bone marrow mononuclear cell administration for acute myocardial infarction patients: The CHINA-AMI randomized controlled trial. Int J Cardiol. 2015 Apr 1;184:446-451. doi: 10.1016/j.ijcard.2015.02.084. Epub 2015 Feb 25. PMID 25755063